CLINICAL TRIAL: NCT00675038
Title: Pilot Study of Non-Invasive Assessment of Hepatic And Myocardial Iron Through T2* MRI In Patients With Iron Overload
Brief Title: Pilot Study of Non-Invasive Assessment of Hepatic And Myocardial Iron Through T2* Magnet Resonance Imaging (MRI) In Patients With Iron Overload
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MRIRON
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Hematological Diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Study participants will be patients who are cared for by the St. Jude Hematology Division and have developed iron overload and require liver biopsy.
  Interventions: Procedure: Liver Biopsy and MRI T2* MRI

INTERVENTIONS:
Procedure: Liver Biopsy and MRI T2* MRI — Evaluation of iron overload with liver biopsy vs. MRI T2* MRI

SUMMARY:
Many hematological disorders are treated by giving red blood cells. Over a long period of time iron from the red blood cell will accumulate in the tissues of the heart, liver, and endocrine glands. This condition is referred to as iron overload and may become life threatening due to the effects of the iron on these tissues. The normal method for evaluation of iron overload is a liver biopsy. This procedure is invasive and has potential risks, such as bleeding and infection.

It is very desirable to establish a method for assessing iron overload which is not invasive. New magnet resonance imaging (MRI) relaxation techniques (T2*MRI) can be used to indirectly assess the liver iron content and iron in the heart. Results of T2*MRIs show excellent correlation with liver iron content and heart function. The use of this method of assessment will minimize the risk and inconvenience of liver biopsy and possibly allow more frequent evaluations for iron overload, thus better treatment for these patients.

Participants in this study will undergo both liver biopsy for liver iron content and T2* MRI of the liver and the heart. Results from the procedures performed in this study will be compared, with the end result being the possible elimination of invasive procedures to diagnose iron overload.

DETAILED DESCRIPTION:
Quantitative measurements of hepatic and cardiac iron by single-breath-hold MRI T2* will allow us to determine the value of this technique as a non-invasive method of monitoring liver and cardiac iron content. By obtaining T2 measurements, we will be able to compare two different techniques for non-invasive iron assessment. With regard to the liver, we will correlate T2* measurements with the gold standard, LIC on liver biopsy. Because it is not feasible to perform cardiac biopsies to evaluate the degree of cardiac hemosiderosis, we will evaluate the relationships between cardiac T2* values and left and right diastolic function, left ventricular ejection fraction, left ventricular end-systolic volume and left ventricular mass index obtained by echocardiography and MUGA scans that are performed as part of the routine clinical care of these patients. In order to estimate whether cardiac T2* values are clinically relevant, we will also investigate the relationship between T2* values and the need for cardiac medication due to cardiac hemosiderosis. Cardiac and hepatic T2* measurements will also be compared to their visual appearances on T2* MR images in order to investigate the relationship between these two assessments. Cardiac and hepatic T2* and their respective visual appearances on T2* MR images will be compared with serum ferritin to evaluate the potential relationships among these measurements of iron overload.

Amen T2* and T2 phantoms are devices that allow calibration of the MR measurements for absolute iron content. Phantoms are test tubes filled with aqueous solutions or gel compounds of materials that mimic various tissue relaxation times (T1, T2 and T2*). Phantoms are commonly used in MRI when quantification is desired. Our phantom will consist of a multitude of small vials which will be visible in the imaging plane. The relaxation times vary in the different vials of the phantom and are known very accurately, especially the T2 and T2* values, which vary over the physiological relevant range. This way the phantom can be used to calibrate the T2* values obtained from the patients heart and liver and eventually be correlated to absolute iron concentrations.

If accurate, the T2* MRI technique would ultimately allow a non-invasive method of quantitatively assessing myocardial and liver iron accumulation, and could predict the degree of morbidity due to iron overload. This new technique could greatly improve the care of our iron overloaded patients by offering a practical and risk free method for evaluation of body iron load. We plan to apply this preliminary information into future studies in this area. Eventually we plan to use the T2* MRI measurements in longitudinal studies of patients with iron overload, both to assess their degree of iron burden and monitor chelation therapy treatments.

Amen Dark blood applications are state-of-the-art in cardiac MRI and commonly applied. There is no risk associated with the dark blood preparation. Comparison of dark and bright blood measurements will show whether both sequences yield similar results and whether one technique is less susceptible to cardiac motion and associated artifacts, thereby offering a higher accuracy and a smaller error in the calculation of T2* and iron concentration.

Information about the heart function can be obtained using MRI techniques, however this information needs to be validated in different populations, such as patients with iron overload. If MR data show a high correlation with echocardiography and MUGA functional data, subsequent protocols could be conducted where the functional information can be gained with an MR measurement, thereby avoid acquiring a MUGA scan and eliminating the exposure to radiation as well as streamlining the protocol by just adding a few additional measurements to an already scheduled MR iron scan. Performing cardiac measurement in a few patients using the MRI technique will allow us to expand the use of this technique for future and larger studies.

Pulmonary hypertension causes progressive right ventricular dysfunction and severe respiratory symptoms (e.g., dyspnea, hypoxemia, poor exercise tolerance, etc.). The association of myocardium iron deposition and its relationship with pulmonary hypertension has not been investigated. Pulmonary hypertension is a prevalent complication among patients with hematologic diseases, especially those with a hemolytic component to the anemia. Because many of these patients are treated with blood transfusion and consequently develop iron accumulation in the heart, the investigation of the association of myocardial hemosiderosis and pulmonary hypertension is warranted.

Finally, because little is understood about iron loading and unloading at the cellular and molecular level, we propose to perform tissue microarray analysis on liver biopsy samples obtained from children with iron overload. This powerful tool will help identify over- and under-expressed genes in the clinical scenario of iron loading, and later in the setting of iron mobilization in these overloaded patients. This pilot study will allow us to investigate differences in gene expression from patients with mild, moderate and severe iron overload, as determined by quantitative LIC on liver biopsy. Our approach will allow characterization of gene expression and analysis for patterns that reflect cellular responses to different degrees of iron overload. This study will not obtain "normal liver" controls from our population, since sickle cell patients without transfusional iron overload have no clinical indication for liver biopsy. It is hoped, however, that subsequent therapeutic protocols will also include microarray studies on liver biopsy samples. In this way, the current microarray analysis will serve as a "baseline" and patients will serve as their own controls for differences in gene expression. This will particularly be important for those patients undergoing successful chelation therapy that should lower LIC. Overall, an understanding of the genetic and biochemical events that regulate these iron loading and unloading processes could greatly improve our ability to treat patients appropriately.

ELIGIBILITY:
Inclusion Criteria:

* Participant is greater than or equal to 7 years of age
* Participant needs a liver biopsy for monitoring iron overload
* Participant is willing to have magnetic resonance testing

Exclusion Criteria:

* Patients with surgical clips placed in the United States after August 15th 1996 will be eligible to participate on the study.
* Contraindication to performing magnetic resonance testing, such as the presence of ferromagnetic material in the body
* Cannot tolerate an MRI without sedation or anesthesia.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinic
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2005-10; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Hankins, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Hankins JS, McCarville MB, Hillenbrand CM, Loeffler RB, Ware RE, Song R, Smeltzer MP, Joshi V. Ventricular diastolic dysfunction in sickle cell anemia is common but not associated with myocardial iron deposition. Pediatr Blood Cancer. 2010 Sep;55(3):495-500. doi: 10.1002/pbc.22587. PMID 20658621
- [Derived] Hankins JS, Smeltzer MP, McCarville MB, Aygun B, Hillenbrand CM, Ware RE, Onciu M. Patterns of liver iron accumulation in patients with sickle cell disease and thalassemia with iron overload. Eur J Haematol. 2010 Jul;85(1):51-7. doi: 10.1111/j.1600-0609.2010.01449.x. Epub 2010 Mar 31. PMID 20374273
- [Derived] Hankins JS, McCarville MB, Loeffler RB, Smeltzer MP, Onciu M, Hoffer FA, Li CS, Wang WC, Ware RE, Hillenbrand CM. R2* magnetic resonance imaging of the liver in patients with iron overload. Blood. 2009 May 14;113(20):4853-5. doi: 10.1182/blood-2008-12-191643. Epub 2009 Mar 4. PMID 19264677
- See also: St. Jude Children's Research Hospital — http://www.stjude.org